CLINICAL TRIAL: NCT04115137
Title: Multicentric Spanish Record of Pelvic Varicose Veins Treated With Vascular Plugs Type Amplatzer - Pelvic Congestion Syndrome: Study of Efficacy and Safety
Brief Title: Pelvic Varicose Veins Treated With Vascular Plugs Type Amplatzer: REPiVAC
Acronym: REPiVAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Group of Research in Minimally Invasive Techniques (Other)
Responsible Party: Sponsor
Other Study IDs: GITMI-05
Record Dates: First submitted 2019-07-11; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Pelvic Congestion Syndrome; Pelvic Varicose Veins; Follow-up Study; Embolization, Therapeutic; Observational Study
Keywords: Pelvic Congestion Syndrome; amplatzer vascular plug; Vascular plug; metallic embolization device; Chronic pelvic pain; embolization procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with pelvic congestion syndrome: Women older than 18 years At least 1 birth Present symptoms
  Interventions: Device: pelvic varicose veins plug embolization

INTERVENTIONS:
Device: pelvic varicose veins plug embolization — pelvic varicose veins plug embolization

SUMMARY:
Spanish multicentric record to study the efficacy and safety of the treatment with plugs in Pelvic Congestion Syndrome.

DETAILED DESCRIPTION:
This is an prospective observational study of patients that have been treated with plugs (type Amplazer) at least one of the pelvic varicose veins.

Patients are recruited when the plug is implanted, and the investigators perfom a patients follow-up during 1, 3, 6, 12, 24 months

ELIGIBILITY:
Inclusion Criteria:

* Female < 18 years
* Present symptomatology
* At least one image diagnosis

Exclusion Criteria:

* Female > 18
* Non present symptomatology
* Non diagnosis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women older than 18, minimun 1 bith
Study Population: Women older than 18 years , minimun 1 bith and with symptoms of pelvic congestion syndrome
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Embolization of pelvic varicose veins using AVP | 24 months
  39/5000 absence of symptoms and vaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A De Gregorio, Ph.D., Principal Investigator — Minimal Invasive Techniques Research Group
Locations (2):
- Spain (2):
  - Lozano Blesa Universitary Hospital, Zaragoza, Aragon
  - Hospital Vithas Nisa Pardo de Aravaca, Madrid

IPD SHARING:
Plan to Share IPD: No